CLINICAL TRIAL: NCT03059966
Title: Evaluation of the Inflammatory and Healing Profile After Root Coverage With Emdogain®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Alexandra Tavares Dias, Researcher, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 285.706
Record Dates: First submitted 2017-01-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enamel Matrix Derivative (Experimental): Microsurgery for root coverage associated with Enamel Matrix Derivative
  Interventions: Biological: Microsurgery technique for root coverage associated to EMD
- Placebo (Placebo Comparator): Microsurgery for root coverage associated with a Placebo comparator
  Interventions: Procedure: Microsurgery technique for root coverage

INTERVENTIONS:
Procedure: Microsurgery technique for root coverage — Microsurgery technique for root coverage adapted for macrosurgery
  Arms: Placebo
Biological: Microsurgery technique for root coverage associated to EMD — Microsurgery technique for root coverage adapted for macrosurgery associated to Enamel Matrix Derivative
  Arms: Enamel Matrix Derivative

SUMMARY:
The purpose of this study was the evaluation of inflammatory and healing profile after root coverage using of Enamel Matrix Derivative. 16 volunteers were selected and submitted to root coverage surgery with subepithelial connective tissue graft, with and without enamel matrix derivative. The patient screening was based in the following inclusion criteria: bilateral recessions in maxillary anterior homologous teeth with aesthetical complaining ou hypersensitivity, non-smokers, healthy and no use of any medication that compromises periodontal health or healing. The split-mouth randomized model was followed in relation to test and control sites. The following clinical parameters were analyzed at baseline and 6-month post-surgery: recession height, recession width, width of keratinized tissue, probing depth, clinical attachment level, and gingival thickness. In addition to the surgical analysis, evaluations of the following inflammatory markers were performed: IL-1β, IL -1RA, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL12, IL-13, IL-15, IL-17, EOTAXIN, FGF, GCSF, GMCSF, IFN-y, IP-10, MCP-1, MIP 1a, PDGF-bb, MIP 1b, RANTES, TNF-α e VEGF. These evaluations were performed at baseline, 7 and 14 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral gingival recessions in homologous teeth

Exclusion Criteria:

* Smokers;
* Systemic diseases;
* Drugs affecting periodontal health/healing.

Ages: 29 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Post-surgical pain | 7 days after surgery
  Questionnaire with a Visual Analog Scale from 0 (no pain) to 10 (worst pain)
Root Coverage Score | 180 days after surgery
  A score including root coverage, marginal gingival tissue contour, mucogingival junction alignment, soft tissue texture and gingival colour according to Cairo et al. (1999)
Post-surgical Clinical Analysis | 180 days after surgery
  Analysis of recession height, recession width, width of keratinized tissue, probing depth, clinical attachment level, and gingival thickness.
Changes in Gingival Fluid Biomarkers | Baseline, 7 and 14 days after surgery
  Analysis for IL-1β, IL -1RA, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL12, IL-13, IL-15, IL-17, EOTAXIN, FGF, GCSF, GMCSF, IFN-y, IP-10, MCP-1, MIP 1a, PDGF-bb, MIP 1b, RANTES, TNF-α e VEGF by Luminex

IPD SHARING:
Plan to Share IPD: No